CLINICAL TRIAL: NCT06101420
Title: Efficacy of Potassium Competitive Acid Blockers (P-CABs) Versus Proton Pump Inhibitors (PPIs) in the First and the Second Lines Eradication Regimens for H. Pylori in Egyptian Patients
Brief Title: Potassium Copetitive Acid Blockers Efficacy in H.Pylori Eradication
Acronym: P-CABs
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Reda Elwakil, Emeritus Professor, Ain Shams University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 111954
Record Dates: First submitted 2023-10-06; First posted 2023-10-26 (Actual); Last update posted 2023-10-26 (Actual); Status verified 2023-10

CONDITIONS: Helicobacter Pylori Eradication
Keywords: P-CABs; Vonoprazan; H.pylori eradication
MeSH Terms: interventions — 1-(5-(2-fluorophenyl)-1-(pyridin-3-ylsulfonyl)-1H-pyrrol-3-yl)-N-methylmethanamine; Clarithromycin; Amoxicillin; Esomeprazole; Levofloxacin; nitazoxanide

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Arm 1 Vonoprazn Triple Therapy Arm (Experimental): Fifty eight participants.The patients received (Clarithromycin 500 mg tablets twice daily[BID]+ Amoxicillin 1gm capsules BID + Vonoprazan 20 mg tablets BID) for 14 days
  Interventions: Drug: Vonoprazan
- Arm 2 Proton Pump Inhibitor Triple Therapy Arm (Active Comparator): Fifty eight participants.The patients received the classic triple therapy (Clarithromycin 500 mg tablets BID + Amoxicillin 1gm capsules BID + Esomeprazole 20 mg tablets BID) for 14 days
  Interventions: Drug: Vonoprazan
- Arm 3 Vonoprazan Quadruple Therapy Arm (Experimental): Fifty eight participants.The patients received a non-bismuth quadruple therapy (Levofloxacin 500 mg tablets once daily[OD] + Vonoprazan 20mg tablets BID + Nitazoxanide 500mg tablets BID +Doxycycline 100mg capsules OD) for 14 days.
  Interventions: Drug: Vonoprazan
- Arm 4 Proton Pump Inhibitor Quadruple Therapy Arm (Active Comparator): Fifty eight participants.The patients received a non-bismuth quadruple therapy (Levofloxacin 500 mg tablets OD + Esomeprazole 20mg tablets BID + Nitazoxanide 500 mg tablets BID +Doxycycline 100mg capsules OD) for 14 days
  Interventions: Drug: Vonoprazan

INTERVENTIONS:
Drug: Vonoprazan — Venoprazan 20mg twice daily,clarithromycin 500mg twice daily,amoxycillin 1 gm twice daily,esomeprazole 20mg twice daily,levofloxacin 500mg a single tablet daily,doxycicline 100mg a single capsule daily and nitazoxanide 500mg twice daily
  Other Names: Clarithromycin; Amoxycillin; Esomeprazole; Levofloxacin; Doxycicline; Nitazoxanide

SUMMARY:
This trial assessed the efficacy of potassium competetor acid blocker (P-CAB) in the eradication of H.pylori

DETAILED DESCRIPTION:
The aim of this study is to compare the effectiveness of Vonaprazan based therapy vs.Proton Pump Inhibitor (PPI)based therapy for the eradication of H.Pylori infection in treatment naive and treatment experienced Egyptian patients.This prospective, non- randomized, controlled study was conducted on symptomatic patients admitted at Tropical Medicine Department at Ain Shams University Hospitals and those presenting at outpatient clinic. The study was conducted in the period from the 1st of January 2022 to the 1st of June 2023.

ELIGIBILITY:
Inclusion Criteria:

* Age above 18 years of both genders.
* Symptomatic patients who has been diagnosed to be H. pylori positive stool by using H. pylori stool antigen test.
* Patients who did not receive H. pylori eradication regimens before were included in group I of the study (First line eradication regimen).
* Patients who received only one eradication regimen before were included in group II of the study (Second line eradication regimen).
* Patients signing an informed consent.

Exclusion Criteria:

* Patients refusing to sign an informed consent.
* Patients who were on PPIs, P-CABs and/or antibiotics starting one month before inclusion in the study .
* Patients who have chronic debilitating and advanced systemic diseases.
* Patients treated with low dose aspirin and/or non-steroidal anti-inflammatory drugs for a long time.
* Any lactating or pregnant female.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 232 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-06-01 (Actual)

PRIMARY OUTCOMES:
H.pylori eradication | six weeks
  The rate of the patients who achieved H.pylori eradication as measured by negative H.Pylori stool antigen test in the four arms of the study was reported.

SECONDARY OUTCOMES:
Safety of Vonoprazan use | six weeks
  The number of patients who reported minor and major treatment connected adverse events in the four arms of the study was reported.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine Ain Shams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No